CLINICAL TRIAL: NCT01250340
Title: Type 2 Diabetes Mellitus: Role of Inflammation and Innate Immunity in The Pathogenesis of Endothelial Dysfunction and Atherosclerosis
Brief Title: Type 2 Diabetes Mellitus and Atherosclerosis
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Roma La Sapienza (Other)
Collaborators: University of Rome Tor Vergata (Other)
Responsible Party: Principal Investigator, Francesco Violi, Full professor of internal medicine, University of Roma La Sapienza
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Diabetes and Oxidative Stress
Record Dates: First submitted 2010-08-30; First posted 2010-11-30 (Estimated); Last update posted 2012-11-28 (Estimated); Status verified 2012-11

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Diabetes; Isoprostanes; Thromboxane; Aspirin
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — Aspirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Aspirin (Experimental): 100 mg/day for 30 days
  Interventions: Drug: Aspirin
- Placebo (Placebo Comparator): 1 cp /day for 30 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Aspirin — 100 mg/day for 30 days
  Arms: Aspirin
Drug: Placebo — 1 cp day for 30 days
  Arms: Placebo

SUMMARY:
In individuals with Type 2 Diabetes (T2D) it has been obtained an outstanding improvement in the management of hyperglycemia, but it has not been achieved a similar result in the reduction of the atherosclerotic syndrome. The comprehension of the mechanisms that link over nutrition to inflammation and innate immune response can be important to understand the relationship between insulin resistance, diabetes mellitus and endothelial dysfunction. It will be investigated: 1) the role of Toll Like Receptors (TLR)s in the pathophysiology of T2D and associated atherosclerosis; 2) the role of aspirin and nicotinamide adenine dinucleotide phosphate (NADPH) oxidase inhibitor/s in the production of TxA2 and F2-isoprostanes in T2D patients; 3)new biomarkers associated to Diabetes and atherosclerosis including markers of endothelial dysfunction and cytokines.

It will be analyzed in isolated platelets from normal controls and/or diabetic patients the production of TxA2, isoprostanes and pro-inflammatory/thrombotic cytokines using aspirin and NADPHoxidase inhibitors.

DETAILED DESCRIPTION:
Study design: prospective, controlled, randomized study. All eligible patients will be randomly assigned in a 1:1 manner to receive aspirin or placebo.

In each recruited subjects we will do:

1. Anamnestic clinical information and Anthropometric measurements
2. Electrocardiogram, echocardiogram and ultrasound assessment of carotid intima-media thickness (IMT) and flow-mediated dilatation (FMD)
3. Ankle-Brachial Index measurement (ABI)
4. blood samples from an antecubital vein after an overnight fast and urine samples at baseline, after 3 days and after 30 days of aspirin (100 mg/day) administration.

Laboratory Methods: Blood samples will be immediately centrifuged at 2,000 rpm for 20 min at 4°C, and the supernatant was collected and stored at -80°C until measurement. All measurements will be done blinded. Samples will be tested in duplicate, and those showing values above the standard curve will be re-tested with appropriate dilutions.Analysis of urinary and platelet isoprostane:Urinary PGF2α-III was measured by a previously described and validated EIA assay method. Ten millilitre urine were extracted on a C-18 SPE column; the purification was tested for recovery by adding a radioactive tracer (tritiated PGF2α-III) (Cayman chemical). The eluates were dried under nitrogen, recovered with 1ml of buffer, and assayed in a PGF2α-III specific EIA kit (Cayman chemical). Urinary PGF2α-III concentration was corrected for recovery and creatinine excretion and expressed as pg/mg of creatinine. PRP was then centrifuged 20 min at 800 g to concentrate platelets and the pellet was suspended in Tyrode buffer to obtain a final platelet concentration of 5x108/mL. PGF2α-III content was measured by a validated EIA assay method as previously described and expressed as pg/mg platelet protein.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 Diabetes Mellitus (defined according to the criteria of the American Diabetes Association)
* Sign of a written informed consent to participate to the interventional study

Exclusion Criteria:

* Liver disease
* Serious renal disorders (serum creatinine >2.5 mg/dL)
* History or evidence of previous major vascular events (myocardial infarction, transient ischemic attack, stroke)
* History of major bleeding
* Autoimmune diseases
* Cancer or present or recent infections
* Use of non-steroidal anti-inflammatory drugs, drugs interfering with cholesterol metabolism, or vitamin supplements or antiplatelet drugs in the previous 30 days

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2010-08; Primary Completion 2011-01 (Actual); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
Changes of isoprostanes after study drug administration. | 3 and 30 days
  Mearuring levels of isoprostanes to understand if isoprostanes could play a crucial role in thrombus formation, independently from Aspirin mediated COX-1 inhibition, supporting their role in the phenomenon of the so call "aspirin resistance" in the setting of T2DM.

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Violi, Study Chair — Divisione di Prima Clinica Medica - Sapienza University of Rome
Locations (1):
- Sapienza Università di Roma, Rome, Italy, Italy

REFERENCES:
- [Derived] Carnevale R, Iuliano L, Nocella C, Bartimoccia S, Trape S, Russo R, Gentile MC, Cangemi R, Loffredo L, Pignatelli P, Violi F; IPINET group. Relationship between platelet and urinary 8-Iso-PGF2alpha levels in subjects with different degrees of NOX2 regulation. J Am Heart Assoc. 2013 Jun 14;2(3):e000198. doi: 10.1161/JAHA.113.000198. PMID 23770972
- [Derived] Cangemi R, Pignatelli P, Carnevale R, Nigro C, Proietti M, Angelico F, Lauro D, Basili S, Violi F. Platelet isoprostane overproduction in diabetic patients treated with aspirin. Diabetes. 2012 Jun;61(6):1626-32. doi: 10.2337/db11-1243. Epub 2012 Mar 16. PMID 22427378